CLINICAL TRIAL: NCT05905809
Title: Controlled, Randomized, Open Label Study to Assess the Efficacy of UniRelieverTM Offloading Brace in the Management of Knee Osteoarthritis
Brief Title: Efficacy of UniRelieverTM Offloading Brace in the Management of Knee Osteoarthritis
Acronym: UNIBRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: MED-RAS GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC43
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Brace; Knee functional capacity; Pain; Compliance
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain; Patient Compliance

STUDY DESIGN:
Intervention Model Description: An interventional, prospective, monocentric, randomized, open and controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I with UniRelieverTM offloading brace (Experimental): Patients wearing the UniRelieverTM offloading brace (THUASNE):
  For intervention group I, in addition to the usual care described above for the control group, patients will wear the studied UniRelieverTM offloading brace.
  Interventions: Device: UniRelieverTM offloading brace (THUASNE)
- Group II with Unloader One® X brace (Experimental): Patients wearing the Unloader One® X brace (Össur):
  For intervention group II, in addition to the usual care described above for the control group, patients will wear the Unloader One® X brace by Össur
  Interventions: Device: Unloader One® X brace (Össur)
- Group III without orthosis (No Intervention): Patients wearing no orthosis:
  In the control group, usual care is defined by:
  * buffer heel and/or
  * insoles and/or
  * outer edge raisin and/or
  * walking stick and/or
  * physiotherapy and/ or
  * analgesics oral and local depending on the patient's needs.

INTERVENTIONS:
Device: UniRelieverTM offloading brace (THUASNE) — The patient will be instructed to wear the brace during walking and physical exercise. The investigator will explain to the patient how to adjust it
  Arms: Group I with UniRelieverTM offloading brace
Device: Unloader One® X brace (Össur) — The patient will be instructed to wear the brace during walking and physical exercise. The investigator will explain to the patient how to adjust it
  Arms: Group II with Unloader One® X brace

SUMMARY:
The objective of this study is to assess the efficacy and performance of a new semi-rigid offloading brace in the management of knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the leading causes of physical disability in the world, affecting a growing portion of the elderly, indeed, it is estimated that 85% of all people over age 60 have some degree of OA.

A survey of 2000 French general practitioners indicated that 10% usually prescribe knee orthoses for patients with knee OA. With the increasing importance of non-pharmacological treatment in recommendations for OA, orthoses will increase in use.

The use of an offloading knee brace that encompasses the knee has proven to be a safe, cost-efficient treatment option for reducing pain and improving function. It can even delay the need for surgery.

The aim of this study is to perform a randomized, prospective, interventional, 3-arm parallel group study to look at the difference in outcome in knee osteoarthritic patient with the use of the new semi-rigid offloading brace versus knee brace comparator versus without orthosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Medial femorotibial knee osteoarthritis grade 2, 3 or 4 according to the Kellgren Lawrence system
* Visual Analog Scale pain ≥ 40/100 in the last 48 hours
* Signed informed consent prior to any study-mandated procedure.
* Affiliated to the General regime of the Social Security or covered by a similar health insurance system

Exclusion Criteria:

* Inability to walk or dependance on a wheelchair or use of crutches.
* Diseases that do not allow participation in the study for a period of six weeks.
* Concomitant ipsilateral patellofemoral osteoarthritis associated with a more severe pain than the one for medial OA.
* Ipsilateral osteoarthritis of the hip associated with a more severe pain than the one for medial OA.
* A body mass index over 35.
* Successful Cortisone injection within the last four weeks before the start of the study.
* Participation to any other clinical study which has an impact on the different endpoints.
* Vulnerable patient, adults being the object of a legal protective measure or enable to express their consent.
* Inability to communicate in German.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Pain-free walking distance | 6 weeks
  The evolution of pain-free walking distance evaluated by reporting the distance that the patient can walk without pain.

SECONDARY OUTCOMES:
Knee functional capacity | 6 weeks
  The evolution of knee functional capacity is evaluated by the Lequesne index completed by the patient at inclusion and six weeks of follow-up (minimum index score 0: None handicap, maximum index score 24: Handicap extremely severe)
Pain on loading | 6 weeks
  The evolution of pain on loading is measured via a numerical rating scale (NRS) after a thirty-minute walk at inclusion and six weeks of follow-up: 0 corresponds to no pain (better outcome) and 10 to maximum pain (worst outcome)
Pain at rest | 6 weeks
  The evolution of pain at rest is measured via a numerical rating scale (NRS) at inclusion and six weeks of follow-up: 0 corresponds to no pain (better outcome) and 10 to maximum pain (worst outcome)
Analgesic consumption | 6 weeks
  The use of analgesics is collected all along the study via a patient's diary completed by the patient every day and via the physician during the inclusion and the six weeks follow-up visit .
Subjective range of movement | 6 weeks
  The subjective knee range of movement is assessed qualitatively by having patients rate it as follow:
  * 'clearly improved',
  * 'improved',
  * 'unchanged',
  * 'deteriorated'
  * 'clearly deteriorated'.
Objective range of movement | 6 weeks
  The objective improvement of knee range of movement is assessed quantitatively by a goniometer (range of movement measure expressed in degrees)
Assessment of Patient's Global Impression of Change (PGI-C) | 6 weeks
  Patient's opinion on Global Impression of Change about his/her general condition by using the PGIC questionnaire completed at the six weeks follow-up visit by the patient. The scale has 7 levels from "no change or condition has got worsed"(worse outcome) to "a great deal better, and a considerable improvement that has made all the difference (better outcome)". Intermediate levels are: "almost the same, hardly any change at all"; "a little better, but no noticeable change", "somewhat better, but the change has not made any real difference"; "moderately better, and a slight but noticeable change"; "better, and a definite improvement that has made a real and worthwhile difference
Assessment of compliance | 6 weeks
  The evaluation of compliance with devices during the duration of the study is reported by the investigator according to the patient's diary completed by the patient each day.
Assessment of patient's satisfaction | 6 weeks
  The evaluation of patient satisfaction with devices is assessed via a self-questionnaire at the end of the study
Assessment of safety (AE and SAEs) | 6 weeks
  The safety of the devices is evaluated by the description of Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring during the study and collected by the patient via the patient's diary and the investigator during follow-up visits:
  * number,
  * type,
  * frequency,
  * intensity,
  * relationship with the study device

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benning, MD, Principal Investigator — Trauma Orthopedic Surgery Practice Center
Locations (1):
- Trauma Orthopedic Surgery Practice Center, Aachen, Friedrich-Wilhelm-Platz 5, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaudreuil J. Orthoses for osteoarthritis: A narrative review. Ann Phys Rehabil Med. 2017 Apr;60(2):102-106. doi: 10.1016/j.rehab.2016.10.005. Epub 2016 Dec 6. PMID 27939833
- [Background] Grazina R, Andrade R, Bastos R, Costa D, Pereira R, Marinhas J, Maestro A, Espregueira-Mendes J. Clinical Management in Early OA. Adv Exp Med Biol. 2018;1059:111-135. doi: 10.1007/978-3-319-76735-2_5. PMID 29736571
- [Background] Hjartarson HF, Toksvig-Larsen S. The clinical effect of an unloader brace on patients with osteoarthritis of the knee, a randomized placebo controlled trial with one year follow up. BMC Musculoskelet Disord. 2018 Sep 22;19(1):341. doi: 10.1186/s12891-018-2256-7. PMID 30243296
- [Background] Maleki M, Arazpour M, Joghtaei M, Hutchins SW, Aboutorabi A, Pouyan A. The effect of knee orthoses on gait parameters in medial knee compartment osteoarthritis: A literature review. Prosthet Orthot Int. 2016 Apr;40(2):193-201. doi: 10.1177/0309364614547411. Epub 2014 Aug 26. PMID 25160784
- [Background] Parween R, Shriram D, Mohan RE, Lee YHD, Subburaj K. Methods for evaluating effects of unloader knee braces on joint health: a review. Biomed Eng Lett. 2019 Jan 23;9(2):153-168. doi: 10.1007/s13534-019-00094-z. eCollection 2019 May. PMID 31168421
- [Background] Petersen W, Ellermann A, Henning J, Nehrer S, Rembitzki IV, Fritz J, Becher C, Albasini A, Zinser W, Laute V, Ruhnau K, Stinus H, Liebau C. Non-operative treatment of unicompartmental osteoarthritis of the knee: a prospective randomized trial with two different braces-ankle-foot orthosis versus knee unloader brace. Arch Orthop Trauma Surg. 2019 Feb;139(2):155-166. doi: 10.1007/s00402-018-3040-8. Epub 2018 Sep 25. PMID 30255369
- [Background] Pham T, van der Heijde D, Altman RD, Anderson JJ, Bellamy N, Hochberg M, Simon L, Strand V, Woodworth T, Dougados M. OMERACT-OARSI initiative: Osteoarthritis Research Society International set of responder criteria for osteoarthritis clinical trials revisited. Osteoarthritis Cartilage. 2004 May;12(5):389-99. doi: 10.1016/j.joca.2004.02.001. PMID 15094138
- [Background] Raja K, Dewan N. Efficacy of knee braces and foot orthoses in conservative management of knee osteoarthritis: a systematic review. Am J Phys Med Rehabil. 2011 Mar;90(3):247-62. doi: 10.1097/PHM.0b013e318206386b. PMID 21273902
- [Derived] Benning M, Villet S, Marques A, Hilgers RD. The effectiveness of the UniReliever offloading knee brace for treating medial knee osteoarthritis: A randomized clinical trial. Prosthet Orthot Int. 2025 Dec 3. doi: 10.1097/PXR.0000000000000503. Online ahead of print. PMID 41331771
- See also: COMMITTEE FOR MEDICINAL PRODUCTS FOR HUMAN USE (CHMP) — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-investigation-medicinal-products-used-treatment-osteoarthritis_en.pdf